CLINICAL TRIAL: NCT01248000
Title: The Use of FDG Positron Emission Tomography (PET)in Patient With Hodgkin Lymphoma (HL) in the "Real World": a Population Based Study From Northern Italy
Brief Title: The Use of FDG-PET in Patient With Hodgkin Lymphoma: a Population Based Study From Northern Italy
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Collaborators: Registro Tumori di Modena (Unknown); Registro Tumori di Reggio Emilia (Unknown); Registro Tumori di Parma (Unknown); registro Tumori di Ferrara (Unknown)
Responsible Party: Massimo Federico, Università di Modena e Reggio Emilia
Other Study IDs: PET-LH
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Histologically Confirmed Classical Hodgkin Lymphoma According to the Current World Health Organisation Classification
Keywords: Hodgkin lymphoma; FDG-PET; prognostic factor; clinical trial
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- classical Hodgkin lymphoma: All cases of classical Hodgkin lymphoma diagnosed between 2006 and 2008 in the province of Modena, Reggio Emilia, Parma and Ferrara will be considered eligible for this study.
  Interventions: Procedure: FDG-PET

INTERVENTIONS:
Procedure: FDG-PET — PET interpretation is based on a site-to-site comparison of FDG uptake both before and after chemotherapy (qualitative approach), according to the criteria defined by Cheson (2008)

SUMMARY:
Positron Emission Tomography (PET) represents a step forward in the definition of response to therapy in patients with Hodgkin Lymphoma (HL). In particular the use of PET for the early assessment of response has been described as the most important tool for predicting the risk of disease progression. As no data are available to support the use of early assessment of response for adapting and modifying subsequent treatment, the use of PET should be limited only to patients enrolled in clinical trials. Irrespective of recommendations PET scanning is included in the current management of patients with HL at baseline, mid treatment, end of treatment, and follow-up. So far no study has been performed to verify how PET is currently used in the clinical setting and to assess if and how results of PET scanning are used for supporting treatment and clinical decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed classical Hodgkin lymphoma according to the current World Health Organisation Classification (nodular sclerosis, mixed cellularity, lymphocyte rich, lymphocyte depleted).
2. Clinical stage I-IV.
3. No previous chemotherapy, radiotherapy or other investigational drug for HL.

Exclusion Criteria:

1. None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases of classical Hodgkin lymphoma diagnosed between 2006 and 2008 in the province of Modena, Reggio Emilia, Parma and Ferrara will be considered eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2009-05; Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | within 1 month after end of treatment
Overall survival | within 1 month after end of treatment
Disease-free survival | within 1 month after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federico, MD, Study Chair — Università di Modena e Reggio Emilia
Locations (1):
- Registro Tumori di Modena, Modena, Modena, Italy